CLINICAL TRIAL: NCT04865042
Title: Short-term Effectiveness of Gabapentin Versus Placebo in Acute Lumbosacral Radiculalgia by Herniation Disc: a Prospective, Multicentric, Randomized, Controlled, Double-blind Study
Brief Title: Short-term Effectiveness of Gabapentin Versus Placebo in Acute Lumbosacral Radiculalgia by Herniation Disc (GRADE)
Acronym: GRADE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC-P0103
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Radiculopathy of Lumbosacral Spine Due to Disc Disorder
Keywords: Radiculalgia; Lumbosacral spine; Disc herniation; Gabapentin
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental): GABAPENTIN per os*:
  * DAY 1:300 mg
  * DAY 2: 600 mg
  * DAY 3: 900 mg
  Interventions: Drug: Gabapentin 300mg
- Placebo (Placebo Comparator): PLACEBO:
  * DAY 1:300 mg
  * DAY 2: 600 mg
  * DAY 3: 900 mg
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Gabapentin 300mg — The patient will receive in addition to the usual analgesic treatment, the treatment under study: Gabapentin.
  During the first 3 days of his hospitalization, an evaluation of the pain and the tolerance to the treatment will be performed.
  The patient will have to take the treatment as follows:
  * Day 1 (1st day of hospitalization): 1 capsule/day
  * Day 2: 2 capsules/day
  * Day 3: 3 capsules/day 72 hours after the first treatment, a blood test will be performed.
  Other Names: NEUROTIN
  Arms: Gabapentin
Drug: PLACEBO — The patient will receive in addition to the usual analgesic treatment, the Placebo During the first 3 days of his hospitalization, an evaluation of the pain and the tolerance to the treatment will be made.
  The patient will have to take the treatment as follows:
  * Day 1 (1st day of hospitalization): 1 capsule/day
  * Day 2: 2 capsules/day
  * Day 3: 3 capsules/day 72 hours after the first treatment, a blood test will be performed.
  Arms: Placebo

SUMMARY:
The study consists in evaluating the analgesic efficacy of Gabapentin versus Placebo in the short term (72h) acute lumbosacral radiculalgia due to disc herniation.

In addition to the usual analgesic treatment, the patient will receive gabapentin or placebo.

During the three days of treatment, an evaluation of the pain and the tolerance will be performed within the two groups: experimental and control.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the analgesic efficacy of GABAPENTIN versus Placebo in 72h for hospitalised patients suffering from acute lumbosacral radiculalgia due to disc herniation.

After signing the consent form, patient's clinical data will be collected and the patient will be allocated to one treatment arm by the randomisation process (ratio 1:1 and stratified on the strong opioid intake).

Two treatment arms are possible :

* Experimental group: GABAPENTINE per os
* DAY1:300 mg
* DAY 2: 600 mg
* DAY3 : 900 mg
* Control group: placebo (same dosage per day as GABAPENTINE).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Radiculalgia or lumboradiculalgia less than 3 months (pain of a lower limb systematized to a radicular territory, possibly associated with lumbar pain),
* Inpatient management for a minimum of 72 hours after inclusion,
* Initial radiculalgia VAS ≥ 4 (moderate to severe pain),
* Concordant disc herniation between clinical symptomatology and imaging (CT or MRI) less than 3 months,
* Written consent signed by the patient,
* Affiliation to a social security system
* For women of childbearing age, use of effective contraception

Exclusion Criteria:

* Motor neurological deficit (≤ 3/5) or cauda equina syndrome (emergency surgical indications),
* Chronic neuropathic pain in the lower limb affected by radiculalgia,
* Lumbar infiltration performed within 72 hours prior to inclusion or unable to be performed after 72 hours,
* Patient already on Gabapentin or Pregabalin, or having taken these treatments in the 7 days prior to inclusion
* Contraindication to Gabapentin (Hypersensitivity to the active substance or to any of the excipients: corn starch, talc, yellow iron oxide, titanium dioxide, sodium lauryl sulfate, gelatin, shellac, propylene glycol, black iron oxide and potassium hydroxide)
* Creatinine clearance < 30ml/min,
* Hemodialysis patient,
* Body weight < 50kgs,
* Transplant patient
* Patient under guardianship or curatorship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analogical Scale (VAS) for radiculalgia | Day 4
  Visual analogue scales are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain being 0 equivalent to no pain and 100 to the worst possible pain between Day 1 (first day) and Day 4, Day 1 corresponding to the first administered dose of the treatment (Gabapentin or Placebo).

SECONDARY OUTCOMES:
Rate of patients with at least one adverse event | Day 7
  Rate of patients with at least one adverse event (all types and grades) between Day 1 and Day 7:
  According to the National Cancer Institute Common terminology criteria for adverse events (NCI CTCAE) v4.0
Change in VAS for lumbalgia | 72 hours
  Change in VAS between Day 1 and Day 4.
Responder rate for lumbalgia at Day 4. | Day 4
  A responder is considered when VAS for low back pain is < 40/100
VAS for radiculalgia | Day 7
VAS for lumbalgia | Day 7
Neuropathic Pain Symptom Inventory (NPSI) scale | Day 7
  The presence of neuropathic pain will be evaluated by the Neuropathic Pain Symptom Inventory (NPSI) scale. This is a self-questionnaire.The tool evaluates mean pain intensity in the last 24h in a verbal numeric scale from zero (no pain) to 10 (worst imaginable pain). Total pain intensity score may be calculated by the sum of 10 descriptors.Evolution of the NPSI (Neuropathic Pain Symptom Inventory) between Day 1 and Day 4, then between Day 1 and Day 7
Dn4 (neuropathic pain screening questionnaire) | Day 7
  In the Dn4 questionnaire there are 4 questions with 10 items. Answers are yes or not. At the end of the questionnaire each "no" is considered as 0, each "yes" is considered as 1. The total score is 10. When addition of answers is 4 or more the test is considered as positive.
Number of interdose of anti-nociceptive analgesics | Day 4
  Number of interdose of anti-nociceptive analgesics between Day 1 and Day 4.
Rate of patients having used at least one interdose | Day 4
  Rate of patients having used at least one interdose between Day 1 and Day 4
Rate of patients having reduced the associated anti-nociceptive analgesic treatment | Day 7
  Rate of patients having reduced the associated anti-nociceptive analgesic treatment (decrease in dosage or step or stop) between Day 4 and and Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ducoulombier, MD, Study Director — GHICL
Locations (5):
- France (5):
  - CH Arras-rheumatology, Arras
  - CH Béthune-rheumatology, Béthune
  - CHU Caen-rheumatology, Caen
  - CH Dunkerque-rheumatology, Dunkirk
  - CHU Rouen-rheumatology, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ducoulombier V, Coquerelle P, Candelier JB, Avenel G, Leroy R, Juilliard A, Norberciak L, Pascart T. Gabapentin versus placebo for the treatment of acute lumbosacral radicular pain caused by disc herniation: study protocol of the GRADE randomized controlled double-blind superiority trial. Trials. 2025 Oct 24;26(1):435. doi: 10.1186/s13063-025-09139-4. PMID 41137125